CLINICAL TRIAL: NCT06462209
Title: Effects of Ladder Training Versus Plyometric Training Program on Agility , Speed and Power in Female Cricket Players
Brief Title: Effects of Ladder Training Versus Plyometric
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0485
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Sports Physical Therapy
Keywords: agility, cricket , ladder training , plyometric
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ladder training (Experimental): ladder training will be given to group 1
  Interventions: Other: ladder training
- plyometric training (Active Comparator): plyometric training will be given to group 2
  Interventions: Other: plyometric training

INTERVENTIONS:
Other: ladder training — Players practiced Ladder training for 60 minutes thrice a week for 8 weeks. There are 3 different types of drills. The first types of drills are steady state drills. These drills focus on quickness Endurance and utilize a constant rhythm throughout the ladder. The second types of drills are burst drills. These drills focus on the ability to turn on rapid burst of foot movement.
  The third types of drills are elastic response drills. These drills focus on improving the reactive speed components of the lower leg. A standard agility ladder is 15 feet long and 20 inches wide Step.
  Arms: ladder training
Other: plyometric training — In plyometric training players practiced for 60 minutes thrice a week for 8 weeks. warm up for 15 minutes , plyometric training for 30 minutes and cool down for 15 minutes
  Arms: plyometric training

SUMMARY:
To determine the effects of ladder training versus plyometric training program on agility, speed and power in domestic female cricket players. Plyometric training program and ladder training program consider effective training methods for players for development of speed, agility and power.

DETAILED DESCRIPTION:
Cricket is a well-known, particularly created team sport that is played on an international scale and involves a group of eleven players. Because both baseball and cricket are played on open fields, they are comparable sports. Cricket was first thought to be a game played only by men.1, 2 However, a few years ago, the globe became aware of the female cricket game because it was becoming more and more popular worldwide. It's a game that requires both physical components and a substantial level of technical understanding. Plyometric and ladder training programmes are thought to be efficient ways to help athletes gain strength, speed, and agility. Players will be selected for this randomised clinical study by use of successive sampling. The players will be split into two groups, 1 and 2, with Group 1 receiving ladder training and Group 2 receiving plyometric training. Each group will receive three 60-minute sessions per week for eight weeks. The vertical leap test, the agility t test, and the 30-dash test will be used to examine patients before and after the trial. Software from SPSS 25 version will be used to analyse the data.

ELIGIBILITY:
Inclusion Criteria:

* • Age ranging from 18-25year.

  * Player with minimum 1- year experience of cricket Only female cricket players.

Exclusion Criteria:

* • Any cardiopulmonary problem. Lower extremity injuries of last 6 months(fractures, ligament ruptures)

  * Players who were unable to complete ladder and plyometric training.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 42 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
vertical jump test | 4 week
  Reaching up with the hand closest to the wall, the athlete stands side by side with the wall. Mark the point of the fingertips this is the standing reach height. The athlete then takes a step back from the wall and launches himself as high while projecting his body upward . At the top of the jump, try to make contact with the wall. The score is the difference in height between the standing reach height and the jump height.
30 dash test | 4 week
  30-yard maximum sprint while timing oneself is part of the exam. Included in the warm-up should be some practice accelerations and starts. The front foot must to land on or behind The tester ought to offer advice on how to run as fast as possible as well as motivation to keep going over the finish line. There can be two trials. If a stopwatch is being used, the time begins at the initial movement.
T test | 4 week
  T test measured both before and after and Athletes can test their agility by running forward, sideways, and backwards in the T-Test. Arrange four cones. At the sound of the timer, the subject begins at cone A, runs to cone B, and places their right hand on the cone's base. Next, they make a left turn, move sideways to cone C, and touch its base with their left hand once more. After that, shuffle sideways to cone D and use your right hand to contact the base. Then they run backwards to cone A and shuffle back to cone B, touching with their left hand.

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young WB, McDowell MH, Scarlett BJ. Specificity of sprint and agility training methods. J Strength Cond Res. 2001 Aug;15(3):315-9. PMID 11710657